CLINICAL TRIAL: NCT03071276
Title: A Phase I/II Study of the Selective Inhibitor of Nuclear Export Selinexor (KPT-330) in Combination With Fludarabine and Cytarabine in Patients With Refractory or Relapsed Leukemia or Myelodysplastic Syndrome
Brief Title: Selinexor in Combination With Fludarabine and Cytarabine in Patients With Refractory or Relapsed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow enrollment
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SELHEM-2; NCI-2014-01704 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Results first posted 2020-04-24 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — selinexor; fludarabine; fludarabine phosphate; Cytarabine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Interventions: Selinexor, Fludarabine, and Cytarabine. Methotrexate/hydrocortisone/cytarabine (intrathecal triples) will be given prior to cycle 1.
  Interventions: Drug: Selinexor; Drug: Fludarabine; Drug: Cytarabine; Drug: methotrexate/hydrocortisone/cytarabine

INTERVENTIONS:
Drug: Selinexor — Given orally on days 1,3,8,10,22 and 24 of each cycle
  Other Names: KPT-330
Drug: Fludarabine — Will be given intravenously (IV) over 30 minutes daily on days 16 through 20. Fludarabine may be given prior to day 16 if it is determined to be in the participant's best interest based on disease progression. Chemotherapy may be delayed by 1-3 days if clinically indicated.
  Other Names: Fludara®; Fludarabine phosphate; 2-fluoro-ara-AMP
Drug: Cytarabine — Will be given IV over 4 hours daily on days 16 through 20. Cytarabine may be given prior to day 16 if it is determined to be in the participant's best interest based on disease progression. Chemotherapy may be delayed by 1-3 days if clinically indicated.
  Other Names: Cytosine arabinoside; Ara-C; Cytosar®
Drug: methotrexate/hydrocortisone/cytarabine — Intrathecal (IT) triples will be given prior to cycle 1: IT cytarabine, IT methotrexate, and IT methotrexate/hydrocortisone/cytarabine (MHA) are acceptable. Patients without evidence of central nervous system (CNS) leukemia will receive no further IT therapy during cycle 1. Patients with CNS disease will receive weekly ITMHA until the cerebrospinal fluid becomes free of leukemia (minimum of 4 doses).
  Other Names: ITMHA; Intrathecal triples

SUMMARY:
This study will be done in two parts: Phase I (NCT02212561) has been completed and published. The goal of the Phase I portion of this study was to find the highest tolerable dose of selinexor (KPT-330) that can be given to patients with leukemia or myelodysplastic syndrome (MDS), when it is combined with fludarabine and cytarabine.

The Phase II portion of the protocol is reflected in this registration.

The goal of the Phase II portion of this protocol is to give the highest dose of selinexor (KPT-330) in combination with fludarabine/cytarabine that was found in Phase I to be safe for children with acute myeloid leukemia (AML). The investigators will examine the effect of this combination treatment.

DETAILED DESCRIPTION:
After the recommended Phase II dose was determined, additional patients began enrolling to receive selinexor at the recommended dose level for further evaluation of tolerability and response.

PRIMARY OBJECTIVE:

* To estimate the overall response rate, as defined by complete response or complete response with incomplete count recovery, of selinexor in combination with fludarabine and cytarabine for patients with relapsed or refractory AML in the phase II portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of AML and must have disease that has relapsed or is refractory to chemotherapy, or that has relapsed after hematopoietic stem cell transplantation (HSCT)

  * Refractory disease is defined as persistent disease after at least two courses of induction chemotherapy.
  * Patients are eligible at first or subsequent relapse or any relapse that is refractory to salvage chemotherapy.
  * Patients must have ≥ 5% leukemic blasts in the bone marrow and/or increasing levels of MRD in the bone marrow as assessed by flow cytometry. If an adequate bone marrow sample cannot be obtained, patients may be enrolled if there is unequivocal evidence of leukemia in the peripheral blood.
* Adequate organ function defined as the following:

  * Direct bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
  * AST (SGOT)/ALT (SGPT) < 3 x IULN
  * Creatinine within normal institutional limits for age
* Prothrombin time (PT) and partial thromboplastin (PTT) ≤ 1.5 x IULN.
* Age criteria: Patients treated at collaborating sites and current St. Jude patients who are on therapy or within 3 years of completion of therapy must be ≤ 24 years old. All other St. Jude patients must be ≤ 21 years old.
* Patients must be able to swallow tablets.
* Performance status: Lansky ≥ 50 for patients who are ≤ 16 years old and Karnofsky ≥ 50% for patients who are > 16 years old.
* Patients must have fully recovered from the acute effects of all prior therapy.
* For patients who have received prior HSCT, there can be no evidence of GVHD and greater than 60 days must have elapsed since the HSCT.

Exclusion Criteria:

* History of cerebellar toxicity or cerebellar neurological findings on exam.
* Must not be pregnant or breastfeeding. Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. For both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose.
* Patients with Down syndrome, acute promyelocytic leukemia, juvenile myelomonocytic leukemia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or other bone marrow failure syndromes are not eligible.
* Use of investigational agents, with the exception of gemtuzumab ozogamicin, within 30 days.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, study participation, follow up, or interpretation of study research.
* Unstable cardiovascular function:

  * symptomatic ischemia
  * congestive heart failure NYHA Class > 3
  * myocardial infarction (MI) within 3 months
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines are acceptable.
* Known human immunodeficiency virus (HIV) infection (pre-study testing not required).
* Patients with malabsorption syndrome, or any other disease significantly affecting gastrointestinal function.
* Prior treatment with selinexor.

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E. Rubnitz, MD,PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (7):
- United States (7):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of Chicago, Chicago, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas

REFERENCES:
- [Result] Alexander TB, Lacayo NJ, Choi JK, Ribeiro RC, Pui CH, Rubnitz JE. Phase I Study of Selinexor, a Selective Inhibitor of Nuclear Export, in Combination With Fludarabine and Cytarabine, in Pediatric Relapsed or Refractory Acute Leukemia. J Clin Oncol. 2016 Dec;34(34):4094-4101. doi: 10.1200/JCO.2016.67.5066. Epub 2016 Oct 31. PMID 27507877
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants must have a diagnosis of AML and must have disease that has relapsed or is refractory to chemotherapy, or that has relapsed after hematopoietic stem cell transplantation (HSCT).
Groups:
- Interventions: Selinexor, Fludarabine, and Cytarabine: Interventions: Selinexor, Fludarabine, and Cytarabine
Period: Overall Study
Arm/Group | Interventions: Selinexor, Fludarabine, and Cytarabine
Started | 37
Completed | 22
Not Completed | 15
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 14

BASELINE CHARACTERISTICS:
Population: Participants must have a diagnosis of AML and must have disease that has relapsed or is refractory to chemotherapy, or that has relapsed after hematopoietic stem cell transplantation (HSCT)
Arm/Group | Interventions: Selinexor, Fludarabine, and Cytarabine
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.65 (6.25)
Age, Continuous [Median (Standard Deviation); unit: years] | 8.04 (6.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: The Overall Response (OR) Rate (Complete Response + Incomplete Count Recovery + Partial Response)
Description: Complete response or complete response with incomplete count recovery or partial response, of selinexor in combination with fludarabine and cytarabine for patients with relapsed or refractory AML in the phase II portion of the study
Time Frame: Between days 28 and 35 of cycle 1 (cycle length is 42-56 days)
Population: Patients with response data available
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interventions: Selinexor, Fludarabine, and Cytarabine
Number analyzed (Participants) | 28
percentage of participants | 53.6 [33.9 to 72.5]

2. Primary Outcome: Complete Response
Description: Complete response, of selinexor in combination with fludarabine and cytarabine for patients with relapsed or refractory AML in the phase II portion of the study
Time Frame: Between days 28 and 35 of cycle 1 (cycle length is 42-56 days)
Population: Patients with response data available
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interventions: Selinexor, Fludarabine, and Cytarabine
Number analyzed (Participants) | 28
percentage of participants | 46.4 [27.5 to 66.1]

3. Primary Outcome: Complete Response or Complete Response With Incomplete Count Recovery
Description: Complete response or complete response with incomplete count recovery, of selinexor in combination with fludarabine and cytarabine for patients with relapsed or refractory AML in the phase II portion of the study
Time Frame: Between days 28 and 35 of cycle 1 (cycle length is 42-56 days)
Population: Patients with response data available
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interventions: Selinexor, Fludarabine, and Cytarabine
Number analyzed (Participants) | 28
percentage of participants | 50.0 [30.6 to 69.4]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected for 30 days after completion of treatment plan or until other anti-leukemia therapy was initiated. If discontinuation from study was due to an AE considered related to study treatment, a follow-up visit was conducted no later than 30 days after the last dose of protocol therapy with recommended safety assessments at least every 30 days, until all toxicities resolved, returned to baseline or became clinically satisfactory, stable, or considered irreversible.
Arm/Group | Interventions: Selinexor, Fludarabine, and Cytarabine
All-Cause Mortality (participants affected / at risk) | 22/37
Serious Adverse Events (participants affected / at risk) | 1/37
Other Adverse Events (participants affected / at risk) | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventions: Selinexor, Fludarabine, and Cytarabine (N=37)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventions: Selinexor, Fludarabine, and Cytarabine (N=37)
Graft Versus host disease (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 30 (133)
Febrile neutropenia (Blood and lymphatic system disorders) | 18 (28)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 4 (6)
Lung infection (Infections and infestations) | 7 (10)
Otitis media (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Soft tissue infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 7 (10)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2)
GGT increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 23 (89)
Neutrophil count decreased (Investigations) | 31 (103)
Platelet count decreased (Investigations) | 33 (360)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 29 (133)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (16)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 11 (41)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 18 (48)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 3 (4)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT03071276/Prot_SAP_000.pdf